CLINICAL TRIAL: NCT03644654
Title: Perioperative Fluid Therapy Optimization in Spinal Surgery Using Non-invasive Measurement of Haemodynamics (ClearSight System, Edwards); a Comparison to Standard Method
Brief Title: Perioperative Fluid Therapy Optimization in Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Principal Investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHospital Hradec Kralove
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hypovolemia; Hypervolemia
Keywords: fluid responsiveness, haemodynamical monitoring, ClearSight
MeSH Terms: conditions — Hypovolemia; Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (Active Comparator): Fluid management will be done according standard care
  Interventions: Procedure: Standard care group
- Noninvasive monitoring group (Experimental): Fluid management will be provided using noninvasive hemodynamical monitor ClearSight (Edwards)
  Interventions: Procedure: Noninvasive monitoring group

INTERVENTIONS:
Procedure: Standard care group — Patient will receive 2 ml/kg/hour of crystalloids (Ringerfundin BBraun) intraoperatively. Fluid boluses will be used according to anesthesiologists decision (timing and amount of fluids). In case of drop of mean arterial pressure (MAP) below 65 mmHg norepinephrine will be started (with initial bolus of 5 - 10 ug).
  Arms: Standard care group
Procedure: Noninvasive monitoring group — Patient will receive 2 ml/kg/hour of crystalloids (Ringerfundin BBraun) intraoperatively. In case of hypotension (defined as a mean arterial pressure below 65 mmHg), the intervention will be led according to a protocol based on cardiac index, systemic vascular resitance and stroke volume variation (SVV) values (ClearSight, Edwards).
  Arms: Noninvasive monitoring group

SUMMARY:
The decision to give fluids perioperatively could be based on methods used to identify preload responsiveness, either invasive or noninvasive estimates of stroke volume variation during mechanical ventilation. This study compares fluid management using continuous noninvasive cardiac output measurement with standard perioperative fluid management.

DETAILED DESCRIPTION:
The aim of the study is to optimise fluid managemet and to reduce perioperative risks during spinal procedures in prone position. Adequate perioperative management guided by hemodynamic monitoring can help to reduce the risk of complications and thus potentially improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma scale 15
* ASA Physical Status Classification System I-III
* planed spinal surgery to 3 hours
* postoperative awakening
* sinus rhythm

Exclusion Criteria:

* NYHA III, IV
* BMI over 40 in females and over 35 in men
* awake operation
* postoperative artificial ventilation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
intraoperative fluid balance | 5 hours
  the difference between fluid intake and output and losses during surgery

SECONDARY OUTCOMES:
mean dose of norepinephrine | 5 hours
  mean dose of norepinephrine wil be calculated as total intraoperative norepinephrine dose devided by the lenght of surgery
level of creatinine | 24 hours
  plasma level of creatinine measured on the first postoperative day
pooperative lung dysfunction | 24 hours
  postoperative lung dysfunction defined as SpO2 value less than 92% or oxygen therapy for more than 6 hours postoperatively
the length of postoperative stay | till 2 months after surgery
  the length of postoperative stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Dostal, MD, Ph.D., Study Director — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

REFERENCES:
- [Result] Kukralova L, Dostalova V, Cihlo M, Kraus J, Dostal P. The Impact of Individualized Hemodynamic Management on Intraoperative Fluid Balance and Hemodynamic Interventions during Spine Surgery in the Prone Position: A Prospective Randomized Trial. Medicina (Kaunas). 2022 Nov 20;58(11):1683. doi: 10.3390/medicina58111683. PMID 36422222